CLINICAL TRIAL: NCT06875388
Title: Effectiveness of Task-specific Training vs Different Yoga Poses With and Without Perturbation to Improve Reactive Balance and Overall Leg Strength in Older Adults
Brief Title: Task-Specific Training vs. Yoga (With and Without Perturbation) for Balance and Leg Strength in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Saima Gul, Associate Professor, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB#545-24
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Functioning of Healthy Individuals; Balance; Strength, Muscle; Quality of Life (QOL)
Keywords: Task-specific training; yoga poses; perturbation; reactive balance; overall leg strength

STUDY DESIGN:
Intervention Model Description: * Appropriate research strategy: Experimental study
  * Appropriate sampling method; non probability convenient sampling
  * Appropriate variable selected & defined; yes
  * State study design; randomized trail
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A: task specific training (Experimental): Group A will receive a basic protocol of 40 minutes involving 10 minutes of warm up 10 10 mins of task-specific training and 10 mins of leg strength exercises and 10 mins of cool-down exercises.
  Interventions: Other: Task specific Training
- Group B specific Yoga poses (Experimental): For group B, a series of yoga poses will be applied. Each training session consists of a 10-minute warm-up, 20 minutes of yoga exercises, and a 10-minute cool-down.
  Interventions: Other: Specific Yoga Poses
- Group C Task specific with perturbation (Experimental): Group C will be 40 minutes involving 10 minutes warm up 10 mins of task-specific training involving perturbation and 10 mins of leg strength exercises involving perturbation and 10 mins of cool-down exercises.
  Interventions: Other: Tasl specific Training with perturbation
- Group D Specific yoga Poses with Perturbation (Experimental): Group D training session consists of a 10-minute warm-up, 20 minutes of yoga exercises with perturbation, and a 10-minute cool-down
  Interventions: Other: Specific yoga poses with perturbation

INTERVENTIONS:
Other: Task specific Training — Group A will receive a basic protocol of 40 minutes involving 10 minutes of warm up 10 10 mins of task-specific training 10 mins of leg strength exercises and 10 mins of cool-down exercises.
  Arms: Group A: task specific training
Other: Specific Yoga Poses — For group B, a series of yoga poses will be applied. Each training session consists of a 10-minute warm-up, 20 minutes of yoga exercises, and a 10-minute cool-down.
  Arms: Group B specific Yoga poses
Other: Tasl specific Training with perturbation — GGroup C will be 40 minutes involving 10 minutes of warm-up 10 minutes of task-specific training involving perturbation 10 mins of leg strength exercises involving perturbation and 10 mins of cool-down exercises.
  Arms: Group C Task specific with perturbation
Other: Specific yoga poses with perturbation — Group D training session consists of a 10-minute warm-up, 20 minutes of yoga exercises with perturbation, and a 10-minute cool-down
  Arms: Group D Specific yoga Poses with Perturbation

SUMMARY:
This experimental study is designed to observe the effectiveness of task-specific training vs yoga with and without perturbation on reactive balance and leg strength in older individuals in Islamabad/Rawalpindi, Pakistan. Older adults meeting the criteria will be grouped into 4 intervention groups. One group will be doing task-specific training, the second will be doing yoga poses, the third will be doing task-specific with perturbation, and 4th will be doing yoga poses with perturbation.

Baseline readings through manual release from lean, minbest test, manual muscle testing (MMT), WHO quality of life, Barthel index, 30-sec sit-to-stand test, Stroop test, and mini-mental state examination, will be taken before starting the intervention, and post-intervention readings will be taken after 3 months of intervention. After this, all readings will be retaken 1 month after stopping the intervention

DETAILED DESCRIPTION:
Plan of Work: males and females above 60 as per eligibility criteria will be enrolled Baseline Assessment: all variables Manual release from leans for reactive Balance, Minbest test questionnaire, Manual Muscle testing, Stroop test, Barthel Index scale, 30 sec-sit to stand test, WHOQOL questionnaire will be measured at the baseline Randomization & Allocation: Eligible consenting subjects will be randomly allocated to all four groups Follow-up Assessment: All the outcome measures observed at baseline will be re-assessed after 3 months of intervention and then 1 month after stopping the intervention.

Statistical Analysis: Pre & post-analysis will be conducted.

study design: it will be an experimental study and non- probability-convenient sampling method will be used. data will be collected from the old homes of Islamabad/ Rawalpindi after seeking approval from the authorities. A randomized control trial will be carried out to enroll older male and female individuals into 4 separate groups with random allocation through the sealed envelope method. 50 individuals will be located in each group. After achieving informed consent from all the participants, a baseline assessment will be conducted. Baseline- and post-intervention assessments of the reactive balance and overall leg strength will be completed one week before the intervention and following the last training session, respectively. Both variables will be tested through reliable tests stated in the next session. Only participants fulfilling the inclusion criteria will be recruited in the study. Then a 12-week intervention of task-specific training vs yoga poses in combination with and without perturbation will be implemented on the study population, having 3 sessions per week and a post-intervention assessment will be conducted afterward

Participants including males and females above 60 will be recruited with no restriction for ethnicity or race. The participants from diverse socio-cultural backgrounds will be considered eligible if they meet the inclusion criteria. The study objective will be explained and participants will be invited to participate based on their free will.

Sampling size: The sample size was calculated using G power and taking the following parameters: Effect size f = 0.25, α err prob = 0.05, Power (1-β err prob) = 0.85, No of groups = 04 Total sample size = 204

Randomization: After assessing the eligibility the participants will be randomly allocated in a study groups through sealed envelop method (group A task-specific training, Group B yoga training, group C task-specific with perturbation, group D yoga with perturbation ). The randomization sequence will done through the sealed envelope method. 200 envelopes will be made ready with the name of each group on 50 envelopes. participants will be asked to pick one envelope. and then their group will be mentioned in the performa.

intervention: Group A will receive a basic protocol of 40 minutes involving 10 minutes warm up 10 10 mins of task-specific training 10 mins of leg strength exercises and 10 mins of cool-down exercises. For group B, a series of yoga poses will be applied. Each training session consists of a 10-minute warm-up, 20 minutes of yoga exercises, and a 10-minute cool-down. Group C will be 40 minutes involving 10 minutes of warm-up 10 mins of task-specific training involving perturbation 10 mins of leg strength exercises involving perturbation and 10 mins of cool-down exercises. Group D training session consists of a 10-minute warm-up, 20 minutes of yoga exercises with perturbation, and a 10-minute cool-down

ELIGIBILITY:
Inclusion Criteria:

* Age above 60
* Males and females with regular medical follow-up, physically autonomous but not doing regular physical activity.
* FRAT Score below 15
* Elders having difficulty in executive function (MMSE score more than 25¬).

Exclusion Criteria:

* • Elderly people confined to bed, using wheelchairs, or unable to walk

  * Elderly individuals with severe cognitive impairment, hemodynamic instability, or severe heart disease.
  * Patients with uncontrolled hypertension, as verified by physicians.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2025-01-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Manual Release from Lean (MRFL) Test: | Outcome measure will be assessed at baseline as a pre-intervention procedure. 2nd time point will be 'immediately after the six-week intervention.' Third time point will be 'through study completion, an average of 3 months
  This methodology assesses balance recovery using MFRL and CRFL-inspired tests. Participants wear a safety harness and stand on a standardized foot placement template (17cm heel distance, 14° angle). Trained personnel and a cushioned mat ensure safety. The test involves a controlled forward lean (≤15°) with sudden release by an administrator. A practice trial familiarizes participants before three test trials. Balance recovery is assessed qualitatively (e.g., stepping, arm use) and quantitatively (distance covered, time). Core muscles, including glutes, hamstrings, and abdominals, stabilize movement. Safety measures include verbal cues, secure harness checks, and moderate perturbations.
Mini Balance Evaluation Systems Test (Mini-BESTest) | Outcome measure will be assessed at baseline as a pre-intervention procedure. 2nd time point will be 'immediately after the six-week intervention.' Third time point will be 'through study completion, an average of 3 months
  The Mini-BESTest is a clinical tool assessing dynamic balance and postural control in individuals with neurological conditions, older adults, and those recovering from injuries. It consists of 14 items across four categories: Anticipatory Postural Adjustments, Reactive Postural Control, Sensory Orientation, and Dynamic Gait. Each item is scored from 0-2, with a maximum score of 28; ≤19 indicates a high fall risk. The test is more sensitive than traditional balance assessments and helps guide rehabilitation by identifying specific impairments and tracking progress. It is widely used in neurology, geriatrics, and rehabilitation for fall prevention and treatment planning.
Manual Muscle Testing (MMT): | Outcome measure will be assessed at baseline as a pre-intervention procedure. 2nd time point will be 'immediately after the six-week intervention.' Third time point will be 'through study completion, an average of 3 months
  Manual Muscle Testing (MMT) is a clinical assessment used to evaluate muscle strength and function by applying resistance against a patient's voluntary movement. It helps diagnose neuromuscular conditions, monitor progress, and guide rehabilitation. MMT grades muscle strength on a 0-5 scale: 0 (no contraction), 1 (visible contraction, no movement), 2 (movement without gravity), 3 (movement against gravity), 4 (movement against moderate resistance), and 5 (normal strength). Testing involves positioning the patient, stabilizing the joint, and applying resistance while observing for compensatory movements. MMT is widely used in physical therapy, neurology, and sports medicine to assess muscular imbalances, nerve injuries, and overall functional capacity. Though subjective, when combined with functional tests and dynamometry, it provides valuable insight into muscle performance, aiding in treatment planning and progress tracking for various musculoskeletal and neurological conditions.
30- secs sit to stand test | Outcome measure will be assessed at baseline as a pre-intervention procedure. 2nd time point will be 'immediately after the six-week intervention.' Third time point will be 'through study completion, an average of 3 months
  The 30-Second Sit-to-Stand Test (30s STS) assesses lower body strength, endurance, and balance, especially in older adults and those with mobility impairments. Participants repeatedly stand from a sturdy chair for 30 seconds, with total repetitions recorded. It evaluates leg strength and functional power, essential for daily activities and fall prevention. Scores ≤12 indicate increased fall risk. Key muscles involved include the quadriceps, gluteus maximus, hamstrings, calves, and core. The test is widely used in clinical and research settings to track rehabilitation progress and guide fall prevention strategies. Its simplicity makes it a reliable tool for identifying mobility decline and designing targeted interventions.
Mini Mental State Examination (MMSE) | Outcome measure will be assessed at baseline as a pre-intervention procedure. 2nd time point will be 'immediately after the six-week intervention.' Third time point will be 'through study completion, an average of 3 months
  used For mental status and cognitive function The Mini-Mental State Examination (MMSE) scores range from 0 to 30, with higher scores indicating better cognitive function; a score of 24 or higher is generally considered normal, while scores below 24 may suggest cognitive impairment.
  Here's a more detailed breakdown of the scoring guide and what the scores mean:
  Scoring:
  Maximum Score: 30 Normal: 24 or higher Mild Cognitive Impairment: 18-23 Moderate Cognitive Impairment: 10-17 Severe Cognitive Impairment: 0-9 <23 is generally accepted as indicating cognitive impairment
  Areas Assessed:
  The MMSE assesses five key areas of cognitive function:
  Orientation: (Time and Place) Registration: (Repeating named prompts) Attention and Calculation: (Serial sevens or spelling "world" backward) Recall: (Registration recall) Language: (Naming a pencil and a watch)

SECONDARY OUTCOMES:
World Health Organization Quality of Life Brief Version ( WHOQOL-BREF ) | Outcome measure will be assessed at baseline as a pre-intervention procedure. 2nd time point will be 'immediately after the six-week intervention.' Third time point will be 'through study completion, an average of 3 months
  For assessing the quality of life:
  1. A shorter, 26-item version of the original 100-item WHOQOL questionnaire. It assesses four domains of quality of life: physical health, psychological health, social relationships, and environment.
  2. It is a self-report questionnaire, meaning individuals answer the questions themselves.
  3. Each of the 26 items in the WHOQOL-BREF is scored on a 5-level scale(e.g., 1- 5), allowing for the calculation of domain-specific and overall quality-of-life scores.
  4. Higher scores generally indicate a better quality of life.
The Barthel Scale/Index (BI) | Outcome measure will be assessed at baseline as a pre-intervention procedure. 2nd time point will be 'immediately after the six-week intervention.' Third time point will be 'through study completion, at an average of 3 months
  Used for assessing functional independence in activities of daily living (ADLs) with scores ranging from 0 to 100 The Barthel Index is a 100-point scale, with each activity assigned a numeric value based on the level of assistance needed.
  Total Score: The total score is calculated by summing the scores for each of the 10 ADLs.
  Higher Scores: Indicate greater independence. Lower Scores: Indicate less independence.
  Interpretation:
  0-20: Total dependency. 21-60: Severe dependency. 61-90: Moderate dependency. 91-99: Slight dependency. 100: Total independence.
Mini Stroop test | Outcome measure will be assessed at baseline as a pre-intervention procedure. 2nd time point will be 'immediately after the six-week intervention.' Third time point will be 'through study completion, at an average of 3 months
  The Mini Stroop Test is a cognitive assessment measuring inhibition, cognitive flexibility, and attentional control. It requires individuals to name the ink color of printed words while ignoring the word itself, assessing the ability to override automatic reading responses. Performance is evaluated based on response time and error rate, with longer times and higher errors indicating cognitive control difficulties. It primarily assesses the prefrontal and anterior cingulate cortex, involved in executive functions like attention and inhibition. Poor performance may indicate issues with cognitive flexibility, inhibitory control, or executive dysfunction seen in ADHD, brain injuries, and frontal lobe disorders. Its simplicity makes it useful in clinical and research settings for identifying cognitive impairments and understanding brain-behavior relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Saima Gul Associate Professor, PhD, Principal Investigator — Shifa Tammer e Millat University, Islamabad, Pakistan
Locations (1):
- Shifa Tameer e Millat University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No